CLINICAL TRIAL: NCT01632579
Title: A Single-Dose, Dose-Escalation Study to Evaluate the Safety and Tolerability of LY3023703 in Healthy Subjects
Brief Title: A Single Dose Study of LY3023703 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 14707; I6H-MC-MCBA (Other: Eli Lilly and Company)
Record Dates: First submitted 2012-06-25; First posted 2012-07-03 (Estimated); Results first posted 2018-08-06 (Actual); Last update posted 2018-08-06 (Actual); Status verified 2018-07

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Celecoxib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Single dose of placebo administered orally on up to one occasion separated by at least a 3 week wash out period.
  Interventions: Drug: Placebo
- LY3023703 (Experimental): Up to 6 single escalating doses of LY3023703 [0.1 milligram (mg) up to 60 mg] administered orally on up to two occasions per participant separated by at least a 3 week wash out period.
  Interventions: Drug: LY3023703
- 400 mg Celecoxib (Active Comparator): Positive control. Single 400 mg dose of celecoxib administered orally, open label, on one occasion separated by at least a 3 week washout period.
  Interventions: Drug: Celecoxib

INTERVENTIONS:
Drug: LY3023703 — Administered orally
  Arms: LY3023703
Drug: Placebo — Administered orally
  Arms: Placebo
Drug: Celecoxib — Administered orally
  Arms: 400 mg Celecoxib

SUMMARY:
This is a phase I study of LY3023703 in healthy participants. The purposes of this study are to look at safety, how well the study drug is tolerated, how much of the study drug gets into the blood stream, and how long it takes the body to get rid of it when given to humans. Information about any side effects that may occur will also be collected. Participants will remain in the study for approximately 3 months. This study is for research purposes only and is not intended to treat any medical condition.

ELIGIBILITY:
Inclusion Criteria:

* Overtly healthy individuals based on the history and physical examinations as determined by the investigator
* Body mass index between 18.5 and 32.0 kilograms per square meter (kg/m^2), inclusive

Exclusion Criteria:

* Have known allergies to LY3023703 or any components of the formulation, celecoxib, or sulfonamides. Participants with known aspirin allergy, allergic reaction to nonsteroidal anti-inflammatory drugs (NSAIDs), or allergies or intolerance to other selective microsomal prostaglandin E synthase (mPGES-1) inhibitors should also be excluded
* Have the presence of active peptic ulcer disease, gastrointestinal (GI) bleeding, chronic gastritis, inflammatory bowel disease, or chronic diarrhea, or positive Helicobacter pylori serology
* Use NSAIDs, celecoxib, aspirin, or acetaminophen (at doses greater than 1 gram per day) within 14 days of screening

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2012-06; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri, 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Evansville, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study had 3 periods. Period 1: 0.1 milligram (mg), 0.5 mg, 2.5 mg LY3023703 or placebo. Period 2: 10 mg, 30 mg, 60 mg LY3023703 or placebo. Period 3: 400 mg celecoxib. There was at least a 3-week washout between periods and at least 7 days between dosing of each cohort in Periods 1 and 2.
Groups:
- Cohort 1 Sequence 1: Participants received LY3023703, placebo and celecoxib capsules orally as per the below dosing sequence in each period.
  Period 1: 0.1 mg LY3023703 in week 1, Period 2: Placebo in week 4 and Period 3: 400mg celecoxib in week 8.
- Cohort 1 Sequence 2: Participants received LY3023703 and celecoxib capsules orally as per the below dosing sequence in each period.
  Period 1: 0.1 mg LY3023703 in week 1, Period 2: 10 mg LY3023703 in week 4 and Period 3: 400mg celecoxib in week 7.
- Cohort 1 Sequence 3: Participants received placebo, LY3023703 and celecoxib capsules orally as per the below dosing sequence in each period.
  Period 1: Placebo in week 1, Period 2: 10 mg LY3023703 in week 4 and Period 3: 400mg celecoxib in week 7.
- Cohort 2 Sequence 1: Participants received LY3023703, placebo and celecoxib capsules orally as per the below dosing sequence in each period.
  Period 1: 0.5 mg LY3023703 in week 2, Period 2: Placebo in week 5 and Period 3: 400mg celecoxib in week 8.
- Cohort 2 Sequence 2: Participants received LY3023703 and celecoxib capsules orally as per the below dosing sequence in each period.
  Period 1: 0.5 mg LY3023703 in week 2, Period 2: 30 mg LY3023703 in week 5 and Period 3: 400mg celecoxib in week 8.
- Cohort 2 Sequence 3: Participants received placebo, LY3023703 and celecoxib capsules orally as per the below dosing sequence in each period.
  Period 1: Placebo in week 2, Period 2: 30 mg LY3023703 in week 5 and Period 3: 400mg celecoxib in week 8.
- Cohort 3 Sequence 1: Participants received LY3023703, placebo and celecoxib capsules orally as per the below dosing sequence in each period.
  Period 1: 2.5 mg LY3023703 in week 3, Period 2: Placebo in week 6 and Period 3: 400mg celecoxib in week 9.
- Cohort 3 Sequence 2: Participants received LY3023703 and celecoxib capsules orally as per the below dosing sequence in each period.
  Period 1: 2.5 mg LY3023703 in week 3, Period 2: 60 mg LY3023703 in week 6 and Period 3: 400mg celecoxib in week 9.
- Cohort 3 Sequence 3: Participants received placebo, LY3023703 and celecoxib capsules orally as per the below dosing sequence in each period.
  Period 1: Placebo in week 3, Period 2: 60 mg LY3023703 in week 6 and Period 3: 400mg celecoxib in week 9.
Period: Period 1 (First Intervention)
Arm/Group | Cohort 1 Sequence 1 | Cohort 1 Sequence 2 | Cohort 1 Sequence 3 | Cohort 2 Sequence 1 | Cohort 2 Sequence 2 | Cohort 2 Sequence 3 | Cohort 3 Sequence 1 | Cohort 3 Sequence 2 | Cohort 3 Sequence 3
Started | 2 | 6 | 2 | 2 | 6 | 2 | 2 | 6 | 2
Received at Least 1 Dose | 2 | 6 | 2 | 2 | 6 | 2 | 2 | 6 | 2
Completed | 2 | 6 | 2 | 2 | 6 | 2 | 2 | 6 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period
Arm/Group | Cohort 1 Sequence 1 | Cohort 1 Sequence 2 | Cohort 1 Sequence 3 | Cohort 2 Sequence 1 | Cohort 2 Sequence 2 | Cohort 2 Sequence 3 | Cohort 3 Sequence 1 | Cohort 3 Sequence 2 | Cohort 3 Sequence 3
Started | 2 | 6 | 2 | 2 | 6 | 2 | 2 | 6 | 2
Completed | 1 | 6 | 2 | 2 | 6 | 2 | 2 | 6 | 2
Not Completed | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 2 (Second Intervention)
Arm/Group | Cohort 1 Sequence 1 | Cohort 1 Sequence 2 | Cohort 1 Sequence 3 | Cohort 2 Sequence 1 | Cohort 2 Sequence 2 | Cohort 2 Sequence 3 | Cohort 3 Sequence 1 | Cohort 3 Sequence 2 | Cohort 3 Sequence 3
Started | 1 | 6 | 2 | 2 | 6 | 2 | 2 | 6 | 2
Received at Least 1 Dose | 1 | 6 | 2 | 2 | 6 | 2 | 2 | 6 | 2
Completed | 0 | 6 | 2 | 2 | 6 | 2 | 2 | 6 | 2
Not Completed | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period
Arm/Group | Cohort 1 Sequence 1 | Cohort 1 Sequence 2 | Cohort 1 Sequence 3 | Cohort 2 Sequence 1 | Cohort 2 Sequence 2 | Cohort 2 Sequence 3 | Cohort 3 Sequence 1 | Cohort 3 Sequence 2 | Cohort 3 Sequence 3
Started | 0 | 6 | 2 | 2 | 6 | 2 | 2 | 6 | 2
Completed | 0 | 6 | 2 | 2 | 6 | 2 | 2 | 6 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 3 (Third Intervention)
Arm/Group | Cohort 1 Sequence 1 | Cohort 1 Sequence 2 | Cohort 1 Sequence 3 | Cohort 2 Sequence 1 | Cohort 2 Sequence 2 | Cohort 2 Sequence 3 | Cohort 3 Sequence 1 | Cohort 3 Sequence 2 | Cohort 3 Sequence 3
Started | 0 | 6 | 2 | 2 | 6 | 2 | 2 | 6 | 2
Received at Least 1 Dose | 0 | 6 | 2 | 2 | 6 | 2 | 2 | 6 | 2
Completed | 0 | 6 | 2 | 2 | 6 | 2 | 2 | 6 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Entire Study Population: Depending on the cohort and period, participants received either an LY3023703 capsule (0.1-mg, 0.5-mg, 2.5-mg, 10-mg, 30-mg, or 60-mg strength) or placebo administered orally once in Periods 1 and 2. In Period 3, participants were administered 400 mg celecoxib, orally. Each dose of study drug was followed by a washout period of at least 3 weeks.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.0 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 29
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 26
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With One or More Drug Related Adverse Events (AEs) or Any Serious AE
Description: AEs that were considered possibly related to study drug, in the opinion of the investigator, were reported. A summary of serious and all other non-serious AEs, regardless of possible study drug relatedness, is located in the Reported Adverse Events module.
Time Frame: Baseline up to Day 7 post-dose
Population: Safety population: participants who received at least 1 dose of study drug or placebo, whether or not he/she completed all the protocol requirements.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Matched placebo capsules administered orally in Periods 1 or 2.
- 0.1 mg LY3023703: 0.1-milligram (mg) LY3023703 capsule administered orally, once in Period 1.
- 0.5 mg LY3023703: 0.5-mg LY3023703 capsule administered orally, once in Period 1.
- 2.5 mg LY3023703: 2.5-mg LY3023703 capsule administered orally, once in Period 1.
- 10 mg LY3023703: 10-mg LY3023703 capsule administered orally, once in Period 2.
- 30 mg LY3023703: 30-mg LY3023703 capsule administered orally, once in Period 2.
- 60 mg LY3023703: 60-mg LY3023703 capsule administered orally, once in Period 2.
- Celecoxib: 400-mg celecoxib dose (two 200-mg celecoxib capsules) administered orally, once in Period 3.
Arm/Group | Placebo | 0.1 mg LY3023703 | 0.5 mg LY3023703 | 2.5 mg LY3023703 | 10 mg LY3023703 | 30 mg LY3023703 | 60 mg LY3023703 | Celecoxib
Number analyzed (Participants) | 12 | 8 | 8 | 8 | 7 | 8 | 8 | 28
Participants
  Any Serious AE | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Drug-Related AE | 3 | 0 | 0 | 0 | 0 | 0 | 1 | 1

2. Secondary Outcome: Pharmacokinetics: Maximum Concentration (Cmax) of LY3023703
Time Frame: Day 1: pre-dose, 0.25, 0.5, 1, 2, 4, 8 and 12 hours, post-dose
Population: Pharmacokinetic (PK) population: participants who received at least 1 dose of study drug and had evaluable Cmax data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | 0.1 mg LY3023703 | 0.5 mg LY3023703 | 2.5 mg LY3023703 | 10 mg LY3023703 | 30 mg LY3023703 | 60 mg LY3023703
Number analyzed (Participants) | 8 | 8 | 8 | 7 | 8 | 8
nanograms per milliliter (ng/mL) | 1.15 (25.4) | 5.66 (27.7) | 23.5 (23.7) | 140 (22.0) | 547 (36.0) | 756 (26.8)

3. Secondary Outcome: Pharmacokinetics: Area Under the Concentration Curve (AUC) of LY3023703
Description: Area under the concentration time curve from the time of dosing to the time of the last observation.
Time Frame: Day 1: pre-dose, 0.25, 0.5, 1, 2, 4, 8 and 12 hours, post-dose
Population: Pharmacokinetic (PK) population: All participants who received at least 1 dose of study drug and had evaluable AUC data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanograms per milliliter (hr*ng/mL)
Arm/Group | 0.1 mg LY3023703 | 0.5 mg LY3023703 | 2.5 mg LY3023703 | 10 mg LY3023703 | 30 mg LY3023703 | 60 mg LY3023703
Number analyzed (Participants) | 8 | 8 | 8 | 7 | 8 | 8
hour*nanograms per milliliter (hr*ng/mL) | 3.19 (52.0) | 54.7 (72.4) | 245 (58.5) | 1680 (36.8) | 9940 (45.6) | 13800 (30.0)

4. Secondary Outcome: Pharmacodynamics: Percent Change From Baseline of ex Vivo Whole Blood Prostaglandin E (PGE) Synthesis After Lipopolysaccharide (LPS) Stimulation
Description: Percent change from baseline of PGE synthesis=(postdose PGE synthesis-baseline PGE synthesis)/baseline PGE synthesis*100, where the unit of measure for PGE synthesis is nanograms per milliliter (ng/ml).
Time Frame: Baseline, 0.5 hours (h), 1 h, 2 h, 8 h, 24 h, and 144 h post-dose
Population: All participants who received at least 1 dose of study drug or placebo and had evaluable PGE data at the specific time points.
Measure: Median (Inter-Quartile Range); unit: percent change in PGE
Arm/Group | Placebo | 0.1 mg LY3023703 | 0.5 mg LY3023703 | 2.5 mg LY3023703 | 10 mg LY3023703 | 30 mg LY3023703 | 60 mg LY3023703 | Celecoxib
Number analyzed (Participants) | 11 | 1 | 8 | 8 | 7 | 8 | 8 | 28
percent change in PGE
  Percent Change at 0.5 h | -10.1 [-36.7 to 71.2] | 102.6 [102.6 to 102.6] | -11.6 [-34.0 to 3.3] | 29.3 [-9.0 to 91.4] | -12.1 [-37.9 to 22.2] | -43.5 [-65.6 to -14.3] | -27.1 [-46.8 to -4.5] | -7.1 [-23.6 to 44.6]
  Percent Change at 1 h | 25.4 [-43.9 to 71.5] | 106.4 [106.4 to 106.4] | -6.2 [-46.4 to 27.3] | -18.9 [-46.8 to 21.8] | -67.6 [-76.9 to -23.8] | -84.1 [-99.8 to -77.7] | -82.4 [-95.1 to -62.1] | -14.0 [-47.1 to 10.5]
  Percent Change at 2 h: number analyzed (Participants) | 11 | 1 | 8 | 8 | 7 | 8 | 8 | 27
  Percent Change at 2 h | 11.2 [-27.1 to 103.2] | 87.9 [87.9 to 87.9] | 52.1 [4.9 to 61.5] | -59.6 [-64.6 to -21.9] | -82.7 [-92.3 to -74.3] | -102.0 [-130.1 to -97.0] | -89.1 [-93.9 to -76.8] | -42.5 [-60.0 to -25.2]
  Percent Change at 8 h: number analyzed (Participants) | 11 | 1 | 8 | 6 | 7 | 8 | 8 | 27
  Percent Change at 8 h | 30.0 [-28.4 to 75.8] | 44.2 [44.2 to 44.2] | 90.5 [76.6 to 113.7] | 3.3 [-16.1 to 40.1] | -56.0 [-81.9 to -52.0] | -96.5 [-111.8 to -94.4] | -96.1 [-100.6 to -87.4] | -26.7 [-42.7 to 6.5]
  Percent Change at 24 h: number analyzed (Participants) | 10 | 0 | 8 | 8 | 7 | 8 | 8 | 27
  Percent Change at 24 h | -29.0 [-47.1 to 8.8] |  | 44.1 [27.5 to 65.0] | -7.6 [-14.7 to 84.1] | 16.1 [-29.9 to 94.4] | -84.2 [-87.1 to -78.1] | -80.7 [-85.6 to -64.2] | -21.8 [-49.9 to 21.0]
  Percent Change at 144 h: number analyzed (Participants) | 11 | 1 | 8 | 8 | 7 | 7 | 8 | 28
  Percent Change at 144 h | -36.8 [-68.0 to -19.4] | -31.1 [-31.1 to -31.1] | 20.5 [-32.0 to 66.6] | 28.9 [-25.3 to 103.9] | 111.6 [66.9 to 117.9] | -61.3 [-115.7 to 68.6] | 4.3 [-21.2 to 36.0] | 11.6 [-28.8 to 190.4]

5. Secondary Outcome: Pharmacodynamics: Percent Change From Baseline of Urinary Excretion of Prostaglandin E(2) Metabolite (PGEM)
Description: Urinary excretion of PGEM, after correcting for urinary creatinine. PGEM was corrected for urinary creatinine by dividing the picograms per milliliter (pg/mL) of metabolite excreted in urine by the concentration of creatinine [milligrams per milliliter (mg/mL)] in urine. Percent change from baseline of urinary excretion of PGEM=(mg creatinine per pg of metabolite excreted in urine postdose-mg of creatinine per pg of metabolite excreted at baseline)/mg of creatinine per pg of metabolite excreted at baseline*100.
Time Frame: Baseline, 0 to 2 hours (h), 2 to 4 h, 4 to 6 h, 6 to 12 h, and 12 to 24 hours post-dose
Population: All participants who received at least 1 dose of study drug or placebo and had evaluable PGEM data at specific time points.
Measure: Median (Inter-Quartile Range); unit: percent change in PGEM
Arm/Group | Placebo | 0.1 mg LY3023703 | 0.5 mg LY3023703 | 2.5 mg LY3023703 | 10 mg LY3023703 | 30 mg LY3023703 | 60 mg LY3023703 | Celecoxib
Number analyzed (Participants) | 12 | 8 | 8 | 8 | 7 | 8 | 7 | 27
percent change in PGEM
  Percent Change at 0 to 2 h: number analyzed (Participants) | 12 | 8 | 7 | 8 | 7 | 8 | 7 | 27
  Percent Change at 0 to 2 h | 4.2 [-26.3 to 30.2] | 7.4 [-35.3 to 14.7] | -4.0 [-19.7 to 19.8] | 1.5 [-15.8 to 17.6] | -5.3 [-21.0 to 47.5] | 17.7 [-24.8 to 35.9] | -6.6 [-25.8 to 52.0] | -7.5 [-28.3 to 11.3]
  Percent Change at 2 to 4 h: number analyzed (Participants) | 12 | 8 | 8 | 8 | 7 | 8 | 7 | 25
  Percent Change at 2 to 4 h | -2.8 [-30.1 to 52.0] | 0.7 [-19.4 to 20.4] | 7.9 [-15.8 to 30.3] | -0.8 [-25.8 to 5.3] | -21.0 [-44.8 to 7.8] | -46.6 [-52.3 to -24.0] | -25.1 [-47.7 to 25.2] | -41.5 [-51.3 to -21.4]
  Percent Change at 4 to 6 h: number analyzed (Participants) | 12 | 7 | 8 | 8 | 6 | 8 | 7 | 25
  Percent Change at 4 to 6 h | -19.0 [-33.7 to 20.6] | -0.0 [-37.8 to 2.9] | -25.0 [-42.4 to -8.9] | -19.0 [-39.7 to -6.7] | -29.1 [-51.6 to -9.0] | -53.0 [-62.5 to -35.7] | -42.4 [-57.3 to 26.9] | -55.0 [-70.3 to -42.6]
  Percent Change at 6 to 12 h: number analyzed (Participants) | 12 | 8 | 7 | 8 | 7 | 8 | 7 | 27
  Percent Change at 6 to 12 h | -18.7 [-45.5 to 11.9] | -18.5 [-36.7 to 7.3] | 2.3 [-31.1 to 10.8] | -20.4 [-27.4 to -7.2] | -39.5 [-57.9 to -23.4] | -37.5 [-62.3 to -19.2] | -48.0 [-58.0 to -9.5] | -49.7 [-68.9 to -27.8]
  Percent Change at 12 to 24 h | -29.7 [-39.3 to 8.6] | -38.8 [-42.1 to -22.9] | -18.0 [-35.8 to 9.2] | -19.1 [-39.9 to -3.5] | -28.8 [-42.6 to 43.3] | -31.2 [-47.7 to -8.6] | -53.0 [-74.9 to -19.9] | -46.2 [-59.2 to -11.4]

6. Secondary Outcome: Pharmacodynamics: Percent Change From Baseline of Urinary Excretion of Prostacyclin Metabolite (PGIM)
Description: Urinary excretion of PGIM, after correcting for urinary creatinine. PGIM was corrected for urinary creatinine by dividing the picograms per milliliter (pg/mL) of metabolite excreted in urine by the concentration of creatinine [milligrams per milliliter (mg/mL)] in urine. Percent change from baseline of urinary excretion of PGIM=(mg creatinine per pg of metabolite excreted in urine postdose-mg of creatinine per pg of metabolite excreted at baseline)/mg of creatinine per pg of metabolite excreted at baseline*100.
Time Frame: Baseline, 0 to 2 hours (h), 2 to 4 h, 4 to 6 h, and 6 to 12 h post-dose
Population: All participants who received at least 1 dose of study drug or placebo and had evaluable PGIM data at specific time points.
Measure: Median (Inter-Quartile Range); unit: percent change in PGIM
Arm/Group | Placebo | 0.1 mg LY3023703 | 0.5 mg LY3023703 | 2.5 mg LY3023703 | 10 mg LY3023703 | 30 mg LY3023703 | 60 mg LY3023703 | Celecoxib
Number analyzed (Participants) | 12 | 8 | 8 | 8 | 7 | 8 | 7 | 27
percent change in PGIM
  Percent Change at 0 to 2 h: number analyzed (Participants) | 12 | 7 | 7 | 8 | 7 | 8 | 7 | 27
  Percent Change at 0 to 2 h | -6.4 [-21.6 to 19.6] | -34.6 [-50.5 to -13.2] | 15.5 [-0.9 to 46.2] | 22.4 [3.5 to 41.9] | -1.2 [-27.3 to 23.7] | 33.1 [-11.9 to 91.1] | 27.7 [-15.6 to 102.0] | -32.0 [-39.2 to -16.2]
  Percent Change at 2 to 4 h: number analyzed (Participants) | 12 | 8 | 8 | 8 | 7 | 8 | 7 | 24
  Percent Change at 2 to 4 h | -10.9 [-34.5 to -2.2] | -19.6 [-34.3 to -13.7] | 18.6 [-18.5 to 49.2] | 9.8 [-3.3 to 64.5] | 29.3 [10.0 to 58.8] | 51.5 [16.3 to 65.6] | 74.5 [-29.6 to 128.2] | -66.0 [-75.9 to -46.5]
  Percent Change at 4 to 6 h: number analyzed (Participants) | 12 | 7 | 8 | 8 | 6 | 8 | 7 | 23
  Percent Change at 4 to 6 h | -0.9 [-29.6 to 29.7] | -19.1 [-58.5 to -5.8] | -3.5 [-13.7 to 11.9] | 3.7 [-17.3 to 23.2] | -0.9 [-27.4 to 36.4] | 19.5 [-2.6 to 67.4] | 63.3 [-18.3 to 138.3] | -60.0 [-68.2 to -53.1]
  Percent Change at 6 to 12 h: number analyzed (Participants) | 12 | 7 | 7 | 8 | 7 | 8 | 7 | 27
  Percent Change at 6 to 12 h | -6.1 [-11.0 to 15.9] | -29.8 [-35.3 to 39.4] | 13.6 [-0.1 to 19.6] | 0.6 [-7.6 to 37.6] | 98.4 [4.9 to 112.3] | 44.1 [14.0 to 98.3] | 49.9 [-10.9 to 138.7] | -45.2 [-57.7 to -23.6]

7. Secondary Outcome: Pharmacodynamics: Percent Change From Baseline of Urinary Excretion of Thromboxane A Metabolite (TXAM)
Description: Urinary excretion of TXAM, after correcting for urinary creatinine. TXAM was corrected for urinary creatinine by dividing the picograms per milliliter (pg/mL) of metabolite excreted in urine by the concentration of creatinine [milligrams per milliliter (mg/mL)] in urine. Percent change from baseline of urinary excretion of TXAM=(mg creatinine per pg of metabolite excreted in urine postdose-mg of creatinine per pg of metabolite excreted at baseline)/mg of creatinine per pg of metabolite excreted at baseline*100.
Time Frame: Baseline, 0 to 2 hours (h), 2 to 4 h, 4 to 6 h, and 6 to 12 h post-dose
Population: All participants who received at least 1 dose of study drug or placebo and had evaluable TXAM data at specific time points.
Measure: Median (Inter-Quartile Range); unit: percent change in TXAM
Arm/Group | Placebo | 0.1 mg LY3023703 | 0.5 mg LY3023703 | 2.5 mg LY3023703 | 10 mg LY3023703 | 30 mg LY3023703 | 60 mg LY3023703 | Celecoxib
Number analyzed (Participants) | 12 | 8 | 8 | 8 | 7 | 8 | 7 | 27
percent change in TXAM
  Percent Change at 0 to 2 h: number analyzed (Participants) | 12 | 8 | 7 | 8 | 7 | 8 | 7 | 27
  Percent Change at 0 to 2 h | -9.1 [-24.2 to 3.4] | -19.9 [-23.6 to -8.4] | 6.5 [-14.1 to 32.4] | -17.9 [-29.7 to -5.8] | 8.7 [-17.2 to 17.0] | 2.7 [-13.4 to 30.4] | -10.2 [-19.8 to -0.1] | -5.0 [-22.5 to 9.8]
  Percent Change at 2 to 4 h: number analyzed (Participants) | 12 | 7 | 8 | 8 | 6 | 8 | 7 | 25
  Percent Change at 2 to 4 h | -12.5 [-23.4 to 3.4] | -11.5 [-25.5 to -3.7] | 11.1 [-4.8 to 23.0] | -7.9 [-23.8 to 2.1] | 21.4 [13.6 to 31.3] | 26.3 [4.1 to 43.1] | 13.0 [-2.3 to 37.3] | -17.7 [-30.8 to -5.9]
  Percent Change at 4 to 6 h: number analyzed (Participants) | 12 | 7 | 8 | 8 | 6 | 8 | 7 | 25
  Percent Change at 4 to 6 h | -15.0 [-21.4 to 2.1] | -19.8 [-24.3 to -5.7] | 2.6 [-4.7 to 12.3] | -18.8 [-20.9 to -13.6] | 16.4 [-1.0 to 32.5] | -13.1 [-25.2 to 7.4] | 18.5 [-3.7 to 22.0] | -25.7 [-37.8 to -18.0]
  Percent Change at 6 to 12 h: number analyzed (Participants) | 12 | 8 | 7 | 8 | 7 | 8 | 7 | 27
  Percent Change at 6 to 12 h | -8.7 [-21.5 to 5.5] | -13.8 [-20.1 to -8.6] | 7.7 [-2.2 to 11.7] | -19.2 [-23.1 to -12.3] | 18.0 [8.7 to 28.8] | 9.8 [-12.1 to 37.7] | 19.1 [14.6 to 31.8] | -16.2 [-26.0 to -4.8]

ADVERSE EVENTS:
Groups:
- LY3023703 0.1 mg: 0.1-milligram (mg) LY3023703 capsule administered orally, once in Period 1.
- LY3023703 0.5 mg: 0.5-mg LY3023703 capsule administered orally, once in Period 1.
- LY3023703 2.5 mg: 2.5-mg LY3023703 capsule administered orally, once in Period 1.
- LY3023703 10 mg: 10-mg LY3023703 capsule administered orally, once in Period 2.
- LY3023703 30 mg: 30-mg LY3023703 capsule administered orally, once in Period 2.
- LY3023703 60 mg: 60-mg LY3023703 capsule administered orally, once in Period 2.
- Celecoxib: 400-mg celecoxib capsule, administered orally, once in Period 3.
Arm/Group | Placebo | LY3023703 0.1 mg | LY3023703 0.5 mg | LY3023703 2.5 mg | LY3023703 10 mg | LY3023703 30 mg | LY3023703 60 mg | Celecoxib
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/8 | 0/8 | 0/8 | 0/7 | 0/8 | 0/8 | 0/28
Other Adverse Events (participants affected / at risk) | 3/12 | 1/8 | 0/8 | 2/8 | 0/7 | 4/8 | 2/8 | 2/28
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=12) | LY3023703 0.1 mg (N=8) | LY3023703 0.5 mg (N=8) | LY3023703 2.5 mg (N=8) | LY3023703 10 mg (N=7) | LY3023703 30 mg (N=8) | LY3023703 60 mg (N=8) | Celecoxib (N=28)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cytomegalovirus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days